CLINICAL TRIAL: NCT02529748
Title: Pilot Study to Assess the Quantitative Dermal Transfer Efficiencies of Solids for Multiple Transfer Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1506M73781
Record Dates: First submitted 2015-08-11; First posted 2015-08-20 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Environmental Exposure
MeSH Terms: interventions — Tinopal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants for Surface Skin Sampling (Experimental): Adult volunteers with healthy, intact skin will have surface skin wipe samples collected following contact with the approved test substances to measure the quantitative transfer of the test substances to and from the skin surface.
  Interventions: Other: Participants for Surface Skin Sampling; Other: Elemental metallic lead; Other: Tinopal

INTERVENTIONS:
Other: Participants for Surface Skin Sampling — Skin wipe samples will be collected to quantify the amount of the test substances transferred to and from the surface of the participants' skin.
  Other Names: No other names
Other: Elemental metallic lead — Consumer product fishing tackle made of elemental lead will be handled by the participants.
  Other Names: No other names
Other: Tinopal — Tinopal, a fluorescent tracer, will be handled by the participants.
  Other Names: No other names

SUMMARY:
Dermal transfer efficiency has been defined as the amount of material that moves from one surface to another following contact. The investigators propose to measure dermal transfer efficiency for the following pathways: (1) object to skin, (2) skin to skin, (3) skin to mouth, (4) clothing to skin, (5) gloves to skin, and (6) air to skin. First, the quantitative dermal transfer will be measured for the two selected test substances (lead, Tinopal) for each of these six pathways. The relative quantities of dermal transfer will also then be compared between the different transfer pathways (e.g., is skin to skin transfer greater or less than clothing to skin transfer?). And second, the pattern of transfer will be characterized semi-quantitatively (e.g., does dermal transfer occur consistently and evenly to the skin from different reservoirs?).

DETAILED DESCRIPTION:
Each of the six transfer pathways will be tested and measured in a controlled, ventilated study chamber at the University of Minnesota's School of Public Health Industrial Hygiene Laboratory. To test each pathway, human volunteers will perform repeated contact activities using an identical protocol (e.g., identical number of contacts, type of material contacted, measured pressure of contact, measured time of contact, measured temperature and humidity) so that inter- and intra-individual variability can be characterized.

The qualitative and quantitative sampling methods that will be used have been developed, tested, and published by researchers from the National Institute for Occupational Safety and Health (NIOSH) and other institutions such as ASTM. Specifically, quantitative transfer efficiencies will be measured using accepted wipe sampling protocols taken from several papers in the peer-reviewed literature. Semi-quantitative transfer patterns will be measured using fluorescent tracer intensity techniques that have also been presented in the peer-reviewed literature. The skin surface wipe samples will be sent to an accredited American Industrial Hygiene Association (AIHA) laboratory for analysis.

These sampling results will allow the investigators to report the measured quantitative dermal transfer efficiencies of elemental metallic lead and Tinopal for each pathway in mass per square surface area of skin, and also calculate the relative transfer efficiencies in terms of percent transferred versus originally loaded. Fluorescent tracer maps will allow the investigators to demonstrate the patterns of transfer for each pathway using intensity of the tracer following transfer. Following this analysis, the investigators will then use the data to better inform the relative importance of the pathways in the conceptual model with respect to dermal exposure assessment and modeling efforts. These results are very important for improving the quality of workplace dermal exposure assessments and techniques. The current approaches are not well validated, and it is unknown if the results of existing dermal exposure models are accurate. It is expected that the results of this study will help to improve the protection of workers from certain dermal exposure hazards in the workplace by providing better inputs to the existing dermal exposure models, since it is not possible to collect exposure samples for each job task in the workplace.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers with healthy intact skin.

Exclusion Criteria:

* Children will be excluded from the study.
* Adults with a past history of dermal sensitization, skin allergy, or dermal irritation or dermatitis because of the potential to have compromised barrier function in the skin.
* Adults who are unwilling to follow protocol requirements.
* Adults who have a documented history of lead poisoning.
* Adults who have a concurrent contagious illness or other stressor which in the opinion of the investigator may interfere with the subject's ability to perform the study's requirements.
* Adults who have open wounds or otherwise compromised skin integrity on their hands.
* Adults who are pregnant or nursing.
* Adults who lack the capacity to provide informed voluntary consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Quantitative mass of test substance per area of skin as measured through surface sampling | Surface samples will be collected within an hour of contact or application
  Participants will handle or touch the approved test substances or an intermediate transfer material such as a solid surface or clothing. Surface skin wipe sampling will then be conducted to measure the amount of material that has been transferred to or from the skin surface.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States